CLINICAL TRIAL: NCT05229575
Title: Breast Stereotactic Radiotherapy to Primary Tumors in Metastatic Patients
Acronym: BoMB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46.20 PAR ComEt CBM
Record Dates: First submitted 2022-01-07; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body Radiation Therapy (SBRT) (Experimental): Patients undergo 5 fractions of image-guided stereotactic body radiation therapy to primary breast tumor over 2 weeks
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Undergo SBRT

SUMMARY:
This is a dose escalation study involving stage IV breast cancer patients not progressing after 6 months of first line systemic treatment. Potential advantages of stereotactic body radiotherapy (SBRT) in treating breast primary tumor in metastatic breast cancer are:

* radio-biological advantage of a short highly effective treatment schedule
* possibility of preventing lesions to become symptomatic
* possibility of continuing systemic treatment without interruption

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Histologically confirmed diagnosis of invasive breast carcinoma (biological immunohistochemical profile: luminal and/or human epidermal growth factor receptor 2 positive)
* Distant metastatic disease not progressing after 6 months of systemic therapy
* Zubrod Performance status of 0-1
* Unifocal tumour < 5 cm tumor size
* Tumor CT or 18-labeled fluorodeoxyglucose positron emission tomography (5FDG-PET) detectable
* No surgery being recommended at time of enrollment.

Exclusion Criteria:

* prior radiotherapy
* active systemic lupus erythematosus, or any history of scleroderma, dermatomyositis with active rash
* Women who are pregnant or lactating.
* Psychiatric or addictive disorders that preclude obtaining informed consent or adherence to protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-10-10 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of stereotactic body radiotherapy (SBRT) | 6 months
  the dose of radiotherapy associated with a ≤ 20% rate pre-specified treatment-related dose -limiting toxicity (DLT) occurring within 6 months from the start of treatment. DLT is defined as any grade 3 or worse toxicity according to CTCAE v.4 related to the following specific symptoms:
  * Radiation dermatitis grade > 3
  * Breast pain grade 3
  * Breast infection grade > 3
  * Breast asymmetry grade 3
  * Fibrosis grade > 3
  * Skin atrophy grade 3
  * Rib fracture grade 3
  * Chest wall pain grade 3

SECONDARY OUTCOMES:
Rate of long-term adverse events | 2 years
  scored according to the NCI CTCAE v. 4.2
Breast Cosmesis | 2 years
  scored according to the European Organization for Research and Treatment of Cancer (EORTC) Cosmetic Rating System for Breast Cancer for the evaluation of cosmetics (score 1 to 4, no difference-large difference by comparing the treated breast to the controlateral breast) and carried out separately by the doctor and the patient
QoL | 2 years
  scored according to the EORTC quality of life questionnaire (QLQ) in breast cancer patients (EORTC QLQ-C30 / BR23)
Primary breast tumor best response | 2 years
  evaluated according to Response Evaluation Criteria in Solid Tumours (RECIST v1.1)

OTHER OUTCOMES:
Primary breast tumor local failure | 2 years
  2 years local failure probability of treated primary tumor predicted by CT planning images

CONTACTS AND LOCATIONS:
Locations (1):
- Università Campus Biomedico, Roma, Italy

REFERENCES:
- [Derived] Ippolito E, Silipigni S, Pantano F, Matteucci P, Carrafiello S, Marrocco M, Alaimo R, Palumbo V, Fiore M, Orsaria P, D'Angelillo RM, Altomare V, Tonini G, Ramella S. BOMB trial: First results of stereotactic radiotherapy to primary breast tumor in metastatic breast cancer patients. Front Oncol. 2023 Mar 17;13:1062355. doi: 10.3389/fonc.2023.1062355. eCollection 2023. PMID 37007063